CLINICAL TRIAL: NCT02182531
Title: Study of the Pharmacokinetic Interactions and Relative Bioavailability of Epinastine and Pseudoephedrine in Healthy Volunteers, Comparing Tablets Containing the Fixed Combination of the Two Substances With Tablets Containing Each of the Two Substances Separately
Brief Title: Epinastine and Pseudoephedrine Fixed Combination Compared to Separate Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 262.255
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — epinastine; Pseudoephedrine

ARMS (3):
- Epinastine and Pseudoephedrine combination (Experimental)
  Interventions: Drug: Epinastine; Drug: Pseudoephedrine; Drug: Epinastine + Pseudoephedrine combination
- Epinastine (Active Comparator)
  Interventions: Drug: Epinastine; Drug: Pseudoephedrine; Drug: Epinastine + Pseudoephedrine combination
- Pseudoephedrine (Active Comparator)
  Interventions: Drug: Epinastine; Drug: Pseudoephedrine; Drug: Epinastine + Pseudoephedrine combination

INTERVENTIONS:
Drug: Epinastine
Drug: Pseudoephedrine
Drug: Epinastine + Pseudoephedrine combination

SUMMARY:
Study to compare the bioavailable fraction of epinastine and pseudoephedrine when administered as a fixed dose combination in tablet form (new pharmaceutical formulation), with that obtained with each of these drugs when administered separately to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes aged between 21 and 45 years
* Non-smoking volunteers
* Volunteers willing to abstain from alcohol
* The volunteers will have to have suspended any drug treatment at least two weeks prior to the start of the study
* Informed consent in writing, signed in time for the start of the study

Exclusion Criteria:

* Women who are pregnant, breast-feeding or receiving hormonal contraceptives
* Volunteers who require drug treatment of any kind of a chronic nature or due to a known addiction
* Volunteers who have taken part in another clinical trial during the preceding four weeks
* Volunteers who have to begin treatment incompatible with this one during the period of the present study (systemic anaesthetics by inhalation, antihypertensives or diuretics used as antihypertensives, beta-adrenergic blockers, CNS (central nervous system) stimulants, digitalis, glycosides, levodopa, monoamine oxidase inhibitors, nitrates, rauwolfia alkaloids, thyroid hormone sympathomimetics)
* Volunteers who do not observe the fasting stipulated in the study or who do not satisfy its requirements with respect to avoiding the ingestion of coffee, tea, cola drinks, etc. during the 24 hours prior to the study
* Volunteers with a history of hepatic or renal disease and disorders of psychiatric origin
* A history of allergy or intolerance with respect to epinastine or pseudoephedrine
* Volunteers who are intolerant of other sympathomimetics (e.g. salbutamol, amphetamine, ephedrine, etc.)
* Non-cooperative volunteers
* Previous participation in this study
* Histories of cardiovascular disease, ischaemic heart disease, hypertension, diabetes mellitus, glaucoma, hyperthyroidism, prostatic hypertrophy

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 1999-08; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the analyte in plasma | Pre-dose, 15, 30, 45 minutes and 1, 2, 4, 6, 8, 12, 24 hours post-dose
Index of the absorption rate Cpmax/AUCt (Peak plasma concentration/Area under the curve from zero to 24 hours) | Pre-dose, 15, 30, 45 minutes and 1, 2, 4, 6, 8, 12, 24 hours post-dose

SECONDARY OUTCOMES:
Peak plasma concentration (Cpmax) | Pre-dose, 15, 30, 45 minutes and 1, 2, 4, 6, 8, 12, 24 hours post-dose
Tmax (Time to reach Cpmax) | Pre-dose, 15, 30, 45 minutes and 1, 2, 4, 6, 8, 12, 24 hours post-dose
T1/2 (Drug half-life) | Pre-dose, 15, 30, 45 minutes and 1, 2, 4, 6, 8, 12, 24 hours post-dose
Number of patients with adverse events | up to 15 days
Number of withdrawals and discontinuations due to safety reasons | up to 15 days
Number of patients with clinically significant changes in vital signs | Baseline, day 1, 8, 15